CLINICAL TRIAL: NCT01655602
Title: Split Wound Comparison of Trichophytic Closure Techniques for Donor Site in Hair Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Assistant Professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SirirajH-005; 825/2554EC3 (Other: SIRB)
Record Dates: First submitted 2012-07-17; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Androgenetic Alopecia
Keywords: Trichophytic closure; hair transplantation; donor site; Androgenetic alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- upper edge trimming (Experimental): Surgery: trichophytic closure The 1-millimetre trimming of upper edge of linear incision before wound closure
  Interventions: Procedure: Trichophytic closure upper edge trimming
- lower edge trimming (Experimental): Surgery: trichophytic closure The 1-millimetre trimming of lower edge of linear incision before wound closure
  Interventions: Procedure: Trichophytic closure lower edge trimming
- Both edge trimming (Experimental): Surgery: trichophytic closure The 0.5-millimetre trimming of both edge of linear incision before wound closure
  Interventions: Procedure: Trichophytic closure both edge trimming

INTERVENTIONS:
Procedure: Trichophytic closure upper edge trimming — 'Trichophytic closure technique' can be done by trimming upper or lower wound edge for about 1 millimeter (as Fig.1) before wound closure. Then the linear scar will be less visible after hair growth. Anyway, there is no exactly wound edge (upper, lower or both) that recommended for the excellent cosmetic results without any severe side effects. Therefore, this study was designed to determine which is the best trichophytic closure technique.
  Other Names: upper Trichophytic; upper edge trimming
  Arms: upper edge trimming
Procedure: Trichophytic closure lower edge trimming — 'Trichophytic closure technique' can be done by trimming upper or lower wound edge for about 1 millimeter (as Fig.1) before wound closure. Then the linear scar will be less visible after hair growth. Anyway, there is no exactly wound edge (upper, lower or both) that recommended for the excellent cosmetic results without any severe side effects. Therefore, this study was designed to determine which is the best trichophytic closure technique.
  Other Names: lower trichophytic closure; lower edge trimming
  Arms: lower edge trimming
Procedure: Trichophytic closure both edge trimming — 'Trichophytic closure technique' can be done by trimming upper and lower wound edge for about 0.5 millimeter (as Fig.1) before wound closure. Then the linear scar will be less visible after hair growth. Anyway, there is no exactly wound edge (upper, lower or both) that recommended for the excellent cosmetic results without any severe side effects. Therefore, this study was designed to determine which is the best trichophytic closure technique.
  Other Names: both edge Trichophytic closure; both edge trimming
  Arms: Both edge trimming

SUMMARY:
This study aim to compare cosmetic results between 3 trichophytic closure techniques for donor site (the trimming of upper, lower and both edge of linear incision) in hair transplantation.

DETAILED DESCRIPTION:
Strip harvesting technique, a conventional hair transplantation procedure, is widely used in the treatment of androgenetic alopecia for more than half a century. It provides less time-consuming, more feasible and more cost-effective comparing with follicular unit extraction (FUE) technique. However, linear scar at the donor site is also introduced.

The latest method to fine the scar at the donor site was invented and known as 'Trichophytic closure technique'. It can be done by trimming upper or lower wound edge for about 1 millimeter (as Fig.1) before wound closure. Then the linear scar will be less visible after hair growth. Anyway, there is no exactly wound edge (upper, lower or both) that recommended for the excellent cosmetic results without any severe side effects. Therefore, this study was designed to determine which is the best trichophytic closure technique.

This research is a pilot, split-wound comparison study of trichophytic closure techniques for donor site in hair transplantation.10 males, aged ≥ 25 years, who require strip harvesting follicular unit transplantation in the treatment of androgenetic alopecia will be enrolled. Preoperative and perioperative process will be conducted as standard procedure except wound closure technique. Each incision wound of donor site will be equally divided into 3 parts (marked with tattoos as Fig.2) and each part will be randomly treated with different trichophytic closure techniques as below.

* The 1-millimetre trimming of upper edge of linear incision before wound closure
* The 1-millimetre trimming of lower edge of linear incision before wound closure
* The 0.5-millimetre trimming of both edge of linear incision before wound closure For evaluation, we have planned to assess both cosmetic results and side effects as shown in the table. ( Table 1 - image file ) After data collecting process, we have planned to analyze the demographic data, rate of infection and other side effects in a descriptive manner. However, the evaluation for cosmetic results will be analyzed by paired t-test in the same technique at different follow up period and by one-way ANOVA between each technique at the same follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age of 25 or more
* Diagnosis of androgenetic alopecia
* Do not response to conventional treatment and undergo hair transplantation surgery

Exclusion Criteria:

* Have skin lesion at donor site
* Psychological disturbance including trichotillomania
* Anti-HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Changing of scar on the donor site during time courses | 1 week, 4 week, 12 week, 24 week
  * Hair density
  * Width of scar
  * Global photographic view (taken with Cannon 60D 18.0 Megapixels 100 mm macro lens)
  * Uninvolved dermatologist's assessment *
  * Self assessment*

SECONDARY OUTCOMES:
Number of Participants with wound complication | immediate, 1week, 4week, 12week, 24week
  Record number of patient who have wound problem example Hematoma, Wound separation, wound Infection, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thuangtong, MD, Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand